CLINICAL TRIAL: NCT00771303
Title: Ruling Out Pulmonary Embolism During Pregnancy:a Multicenter Outcome Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Collaborators: Swiss National Science Foundation (Other); University Hospital, Brest (Other)
Responsible Party: Principal Investigator, Marc Righini, Prof, University Hospital, Geneva
Other Study IDs: 3200B0-120760; Swiss medical Foundation
Record Dates: First submitted 2008-10-10; First posted 2008-10-13 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Pulmonary Embolism; Deep Vein Thrombosis
Keywords: Pregnancy; Pulmonary embolism; MSCT
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis | interventions — fibrin fragment D

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Nt-pro BNP measurement
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Ct scan: Pregnant patients with suspected PE will undergo a strategy based on clinical probability assessment, D-dimer measurement, lower limb compression ultrasonography and multi-slice computed tomography.
  Interventions: Other: Pregnant patients with suspected PE will undergo a strategy based on clinical probability assessment, D-dimer, lower limb vein ultrasonography and MSCT.

INTERVENTIONS:
Other: Pregnant patients with suspected PE will undergo a strategy based on clinical probability assessment, D-dimer, lower limb vein ultrasonography and MSCT.

SUMMARY:
Venous thromboembolism (VTE) remains a major cause of maternal morbidity and mortality in developed countries. Objective diagnosis of pulmonary embolism (PE) and/or deep vein thrombosis (DVT) in pregnancy is crucial. Failure to identify PE or/or DVT will place the mother's life at risk, and unnecessary treatment will not only expose her to anticoagulants but will also label her as having had VTE. Thus, this diagnosis has serious implications for the management of her present pregnancy, and for other aspects of her life ranging from contraception to thromboprophylaxis in future pregnancies and hormone replacement therapy in later life. It is therefore critical that all women with symptoms or signs that suggest venous thromboembolism have appropriate investigation and diagnosis based on objective diagnostic tests.

The current diagnostic approach in suspected PE is based on sequential diagnostic tests: 1) assessment of clinical probability, 2) fibrin D-dimer measurement, 3) compression ultrasonography of lower limb veins and 4) multi-slice computed tomography (MSCT). However, physicians are reluctant to perform MSCT in pregnant women because of potential adverse effect of radiation exposure to the fetus. For this reason, ventilation/perfusion or perfusion-only lung scan has been the cornerstone of PE diagnosis in pregnant women. Indeed, perfusion lung scan was assumed to be associated with less radiation than computed tomography (CT). However, this technique is now widely abandoned in the usual diagnostic strategy of PE for the following reasons: it is not widely available; its interpretation may be difficult and the test may be inconclusive in the presence of other chest abnormalities. Moreover, recent data convincingly show that the radiation exposure associated with single-slice or multi-slice CT exposes the fetus to less radiation than perfusion lung scan.

However, the use of CT has never been adequately validated in pregnant women with clinically suspected PE. The investigators, therefore, plan to set up a prospective management study in which pregnant women with suspected PE will undergo a sequential diagnostic strategy based on 1) assessment of clinical probability 2) D-dimer measurement 3) compression ultrasonography, and 4) MSCT.

Nowadays, the overestimated fear of radiation exposure for the fetus leads to an irrational attitude and inadequate investigations in pregnant women with suspected PE, even though both European [3, 4] and North-American guidelines [5] suggest that only objective testing may accurately rule out the disease. The proposed study should lead to an increased awareness of the risks and benefits of appropriate imaging in pregnant women suspected of PE and should result in a more rational management of this under-studied patient group.

DETAILED DESCRIPTION:
Venous thromboembolism (VTE) remains a major cause of maternal morbidity and mortality in developed countries. Objective diagnosis of pulmonary embolism (PE) and/or deep vein thrombosis (DVT) in pregnancy is crucial. Failure to identify PE or/or DVT will place the mother's life at risk, and unnecessary treatment will not only expose her to anticoagulants but will also label her as having had VTE. Thus, this diagnosis has serious implications for the management of her present pregnancy, and for other aspects of her life ranging from contraception to thromboprophylaxis in future pregnancies and hormone replacement therapy in later life. It is therefore critical that all women with symptoms or signs that suggest venous thromboembolism have appropriate investigation and diagnosis based on objective diagnostic tests.

Diagnosis of VTE on a clinical basis is unreliable, especially during pregnancy because leg swelling and mild dyspnea are frequent during normal pregnancy.

The current diagnostic approach in suspected PE is based on sequential diagnostic tests: 1) assessment of clinical probability, 2) fibrin D-dimer measurement, 3) compression ultrasonography of lower limb veins and 4) multi-slice computed tomography (MSCT). However, physicians are reluctant to perform MSCT in pregnant women because of potential adverse effect of radiation exposure to the fetus. For this reason, ventilation/perfusion or perfusion-only lung scan has been the cornerstone of PE diagnosis in pregnant women. Indeed, perfusion lung scan was assumed to be associated with less radiation than computed tomography (CT). However, this technique is now widely abandoned in the usual diagnostic strategy of PE for the following reasons: it is not widely available; its interpretation may be difficult and the test may be inconclusive in the presence of other chest abnormalities. Moreover, recent data convincingly show that the radiation exposure associated with single-slice or multi-slice CT exposes the fetus to less radiation than perfusion lung scan.

However, the use of CT has never been adequately validated in pregnant women with clinically suspected PE. We, therefore, plan to set up a prospective management study in which pregnant women with suspected PE will undergo a sequential diagnostic strategy based on 1) assessment of clinical probability 2) D-dimer measurement 3) compression ultrasonography, and 4) MSCT.

Nowadays, the overestimated fear of radiation exposure for the fetus leads to an irrational attitude and inadequate investigations in pregnant women with suspected PE, even though both European and North-American guidelines suggest that only objective testing may accurately rule out the disease. The proposed study should lead to an increased awareness of the risks and benefits of appropriate imaging in pregnant women suspected of PE and should result in a more rational management of this under-studied patient group.

ELIGIBILITY:
Inclusion Criteria:

* All pregnant patients with a clinical suspicion of acute PE will be included in the study, provided they correspond to the following diagnostic and exclusion criteria, and they have signed an informed consent form.

Exclusion Criteria:

* Age less than 18 years
* Absence of informed consent
* Patients allergic to contrast medium
* Impaired renal function (creatine clearance less than 30 ml/min as estimated by the Cockroft formula)
* Geographic inaccessibility for follow-up

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with suspected PE.
Sampling Method: Non-Probability Sample
Enrollment: 402 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with a symptomatic thromboembolic event in the three month follow-up among those in whom PE was ruled out by the diagnostic strategy and who were left untreated by anticoagulants. | 3 months

SECONDARY OUTCOMES:
Efficacy of non invasive testing | 3 months
Proportion of patients with a negative D-dimer result | 3 months
Proportion of patients with a lower limb venous ultrasound showing a proximal DVT | 3 months

CONTACTS AND LOCATIONS:
Locations (9):
- France (8):
  - Pierre-Marie ROY, Angers
  - Grégoire LE GAL, Brest
  - Florence PARENT, Clamart
  - Isabelle QUERE, Montpellier
  - Jean-Christophe GRIS, Nîmes
  - Guy MEYER, Paris
  - Caroline BOHEC, Pau
  - Antoine ELIAS, Toulon
- Marc Righini, Geneva, Switzerland